CLINICAL TRIAL: NCT01279434
Title: Vitamin E Versus Vitamin E Plus Pentoxiphyllin in Patients With Nonalcoholic Steatohepatitis: A Prospective Randomized Clinical Trial
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Sponsor: Institute of Liver and Biliary Sciences, India (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ILBS/DHPT/CT/006
Record Dates: First submitted 2010-12-25; First posted 2011-01-19 (Estimated); Last update posted 2015-05-28 (Estimated); Status verified 2011-11

CONDITIONS: Non Alcoholic Steatohepatitis
MeSH Terms: conditions — Non-alcoholic Fatty Liver Disease | interventions — Vitamin E

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Vitamin E plus Pentoxiphyllin (Experimental)
  Interventions: Drug: Vitamin E plus Pentoxiphyllin
- Vitamin E (Active Comparator)
  Interventions: Drug: Vitamin E

INTERVENTIONS:
Drug: Vitamin E plus Pentoxiphyllin — Both drugs will be administered daily Vit E (400 mg BD) and pentoxiphyllin (400 mg TDS) for 12 months
  Other Names: Arm A
  Arms: Vitamin E plus Pentoxiphyllin
Drug: Vitamin E — Vitamin E 400 mg BD daily for 12 months
  Other Names: Arm B
  Arms: Vitamin E

SUMMARY:
Nonalcoholic fatty liver disease (NAFLD) is a spectrum of hepatic pathology, ranging from simple steatosis, steatohepatitis, to cirrhosis. Nonalcoholic steatohepatitis (NASH) is a more advanced form of disease where steatosis is accompanied by hepatocyte injury as well as infiltration of inflammatory cells. Since, both vitamin E and PTX has been found to improve NASH when used alone, a combination of these two should be expected to give better results because of targeting two different pathogenetic mechanisms (cytokines amplification and oxidative stress) in NASH patients. This will be open labelled, prospective, randomized study. The diagnosis of NAFLD will be made on the basis of Ultrasonographic findings suggestive of fatty liver and presence of insulin resistance or features of metabolic syndrome. Subsequently histologic confirmation of the diagnosis of NASH will be made in all cases.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of NAFLD by ultrasonographic
* Presence of Insulin resistance
* Histological confirmation of NASH
* Increased transaminases (>1.5 upper limit normal [ULN])

Exclusion Criteria:

* Patients with alcohol > 20g/ day
* Other known liver disease
* Medications known to induce fatty liver

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2012-01; Primary Completion 2012-03 (Estimated); Study Completion 2012-06 (Estimated)

PRIMARY OUTCOMES:
Improvement in hepatocyte injury and fibrosis (NAFLD Activity Score [NAS score]) | Baseline and 1 year

SECONDARY OUTCOMES:
Normalization of serum transaminases levels | Baseline and 1 year
Reduction in serum levels of proinflammatory cytokines (TNF-α and IL-6) and Malondialdehyde (MDA). | Baseline and 1 year
Improvement in HOMA-IR | Baseline and 1 year
No worsening of fibrosis | Baseline and 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Dr Ramesh Kumar, MD,DM, Principal Investigator — Institute of Liver and Biliary Sciences
Locations (1):
- Institute of Liver & Biliary Sciences, New Delhi, National Capital Territory of Delhi, India